CLINICAL TRIAL: NCT00711555
Title: An Open Label Phase II Study of Aprepitant for Multi-day Moderately-high to Highly Emetogenic Chemotherapy Regimens
Brief Title: Emend for Multiple-day Emetogenic Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stacy Shifflett Shord, Assistant Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-0363; NCT00229489 (obsolete NCT alias)
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Nausea; Vomiting
Keywords: nausea; vomiting; multiple days; chemotherapy; serotonin receptor antagonist; corticosteroids; aprepitant; rescue therapy
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant; Ondansetron; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm study with Emend (Experimental): On day 1, the subject will receive a total daily dose of oral dexamethasone 12mg, oral ondansetron 24mg, and oral aprepitant 125mg. On days 2 to THE LAST DAY OF THE MODERATELY-HIGH TO HIGHLY EMETOGENIC CHEMOTHERAPY, subjects will receive a total daily dose of oral dexamethasone 12mg, oral ondansetron 24mg, and oral aprepitant 80mg. All anti-emetics should be give one hour before starting chemotherapy administration.
  FOR TWO DAYS AFTER RECEIVING CHEMOTHERAPY, the subject will be prescribed oral dexamethasone 4mg every 12 hours and oral aprepitant 80 mg every day.
  Interventions: Drug: aprepitant, ondansetron, dexamethasone

INTERVENTIONS:
Drug: aprepitant, ondansetron, dexamethasone — On day 1, the subject will receive a total daily dose of oral dexamethasone 12mg, oral ondansetron 24mg, and oral aprepitant 125mg. On days 2 to THE LAST DAY OF THE MODERATELY-HIGH TO HIGHLY EMETOGENIC CHEMOTHERAPY, subjects will receive a total daily dose of oral dexamethasone 12mg, oral ondansetron 24mg, and oral aprepitant 80mg. All anti-emetics should be give one hour before starting chemotherapy administration.
  FOR TWO DAYS AFTER RECEIVING CHEMOTHERAPY, the subject will be prescribed oral dexamethasone 4mg every 12 hours and oral aprepitant 80 mg every day.
  FOR RESCUE, the subject will be prescribed prochlorperazine 10 mg oral every 4 hours as needed for nausea and prochlorperazine 10 mg intravenous every 4 hours as needed for vomiting.

SUMMARY:
The purpose of the study is to assess the effect of Emend (aprepitant) on nausea and vomiting associated with chemotherapy. Chemotherapy commonly causes nausea and vomiting and this affects patients' quality of life and attitudes toward treatment. Although nausea and vomiting associated with chemotherapy has been decreasing due to improved therapy, some patients will still experience this side effect. Therefore, new medications are needed to decrease the amount of nausea and vomiting patients have with chemotherapy. Emend (aprepitant) is a new medication used to treat nausea and vomiting with chemotherapy, but it has only been studied in patients receiving only one dose of chemotherapy that makes most people sick. However, there is little experience with this medication in patients receiving multiple days of chemotherapy that causes nausea and vomiting.

DETAILED DESCRIPTION:
In the studies leading to aprepitant's approval, subjects received only one dose of highly emetogenic chemotherapy. Campos et al studied subjects who received their first course of cisplatin containing chemotherapy that included a cisplatin dose 70mg/m2 and reported that aprepitant in addition to granisetron and dexamethasone increased the number of subjects without acute or delayed emesis (p<0.01). A similar study done by Poli-Bigelli et al indicated that adding aprepitant to a standard antiemetic regimen increased the percentage of subjects without emesis and using rescue therapy during the acute phase (83% to 69%; p < 0.001). Adding aprepitant also increased the percentage of subjects with no emesis or use of rescue medications in the delayed phase (68% vs. 47%, p<0.001). Although these studies demonstrate the benefits of aprepitant for a one day chemotherapy regimen, the benefits of adding aprepitant to current standard antiemetic therapy (dexamethasone plus a serotonin receptor antagonist) in subjects receiving multiple days of moderately-high to highly emetogenic chemotherapy have not been examined within a clinical study. We hypothesize that aprepitant with dexamethasone and a serotonin receptor antagonist from days one to two days after finishing chemotherapy will decrease nausea for subjects receiving chemotherapy regimens that include multiple days of treatment with moderately-high to highly emetogenic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a life expectancy > 3 months
* Subjects with an ECOG performance score < 3
* Subjects with access to a telephone for follow-up
* Subjects able to swallow tablets and capsules

Exclusion Criteria:

* Subjects who previously received aprepitant as prophylaxis for chemotherapy induced nausea and vomiting.
* Subjects with an allergy, hypersensitivity, or contraindication to aprepitant, dexamethasone, prochlorperazine or a serotonin receptor antagonist.
* Subject with uncontrolled diabetes or a concurrent illness/condition requiring chronic systemic steroids or pre-existing gastrointestinal pathology.
* Subjects with a history of excessive alcohol consumption.
* Women who are pregnant or lactating.
* Subjects with nausea at baseline or chronically using other antiemetic agent(s).
* Subjects currently receiving another investigational agent.
* Subjects taking a medication that can interact with aprepitant, including the following medications:

  * warfarin
  * oral contraceptives
  * tolbutamide
  * phenytoin
  * midazolam
  * ketoconazole
  * rifampin
  * paroxetine
  * diltiazem
* Subjects with poor hepatic or renal function defined as AST > 3 x ULN, ALT > 3 x ULN, total bilirubin > 3 x ULN, alkaline phosphatase > 3 x ULN or serum creatinine >2 mg/dl measured within three months before starting chemotherapy.

Subjects with hepatic metastases with AST > 5 x ULN, ALT > 5 x ULN, total bilirubin > 5 x ULN, alkaline phosphatase > 5 x ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Shord, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Started | 22
Completed | 19
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (Percentage of Patients)
Description: defined as a no emetic episodes and no use of rescue therapy
Time Frame: cycle 1, day 1
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 19
percentage of participants | 84

2. Secondary Outcome: Complete Protection
Description: defined as no emesis, no use of rescue medications, and a maximum nausea severity < 25 mm (100 mm visual analog scale, 0 = no nausea, 100 = worst nausea)
Time Frame: cycle 1, day 1
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 19
percentage of participants | 74

3. Secondary Outcome: no Emesis
Time Frame: cycle 1, day 1
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 19
percentage of participants | 100

4. Secondary Outcome: no Nausea
Description: defined as maximum nausea severity < 5 mm (100 mm visual analog scale, 0 = no nausea, 100 = worst nausea)
Time Frame: cycle 1, day 1
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 19
percentage of participants | 74

5. Secondary Outcome: no Significant Nausea
Description: defined as a maximum nausea severity < 25 mm (100 mm visual analog scale, 0 = no nausea, 100 = worst nausea)
Time Frame: cycle 1, day 1
Measure: Number; unit: percentage of participants
Arm/Group | Aprepitant, Dexamethasone, Ondansetron, Multiple Days
Number analyzed (Participants) | 19
percentage of participants | 79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes